CLINICAL TRIAL: NCT03325166
Title: The Use of Perfusion MRI Using Ferumoxytol and Small Molecular Weight Gadolinium (Gd) Agents to Assess Response to Pembrolizumab in Brain Metastases and Systemic Lesions in NSCLC: A Comparison of Imaging Modalities to Address Brain Metastases, Pseudoprogression, and Systemic Lesion Tumor Flare (Neuro-Check Pilot)
Brief Title: Pembrolizumab and Magnetic Resonance Imaging With Ferumoxytol in Treating Patients With Non-small Cell Lung Cancer and Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016709; NCI-2017-01730 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016709 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-10-06; First posted 2017-10-30 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Lung Carcinoma Metastatic in the Brain; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, ferumoxytol MRI) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (or up to 32 cycles) in the absence of disease progression or unacceptable toxicity. Patients also receive ferumoxytol IV and undergo MRI at baseline, 12 weeks after radiation, at suspected radiographic progression, and 6 weeks after suspected radiographic progression.
  Interventions: Drug: Ferumoxytol; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This pilot phase II trial study evaluates the usefulness of the ferumoxytol steady state magnetic resonance imaging (MRI) technique for response assessment after pembrolizumab and radiation therapy in non-small cell lung cancer that has spread to the brain (brain metastases). The interactions of monoclonal antibodies such as pembrolizumab, and the body's immune system may result in an anti-tumor effect. However, it may also increase inflammation around the tumor which cannot be differentiated from true tumor growth on standard MRI. This study evaluates ferumoxytol as an MRI contrast agent to differentiate this treatment related inflammation from true tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the sensitivity and specificity of relative cerebral blood volume (rCBV) measured by steady state magnetic resonance imaging (MRI) with ferumoxytol in predicting true versus (vs) pseudoprogression after stereotactic radiosurgery (SRS) and intravenous (IV) pembrolizumab in subjects with brain metastases from non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. Evaluate the safety and tolerability of pembrolizumab when given with SRS in subjects with brain metastasis.

II. Evaluate progression free survival, overall survival, best response in brain disease, best response in systemic disease, and duration of best responses of brain and systematic diseases.

EXPLORATORY OBJECTIVES:

I. Compare the immune response as determined by the volume, pattern and intensity of delayed (24 hour [hr]) ferumoxytol uptake between subjects who develop true vs pseudoprogression.

II. Investigate the serum immunological parameters and correlate clinical as well as radiological response with systemic immune response to pembrolizumab as measured by immunological panel.

III. Compare the changes percentage expression in PDL-1 in the biopsy tissue before and after therapy at the time of progression.

IV. In subjects with measurable systemic lesions, investigate the feasibility of measuring vascular volume fraction (VVF), vessel size index (VSI) and vessel density index (VDI) as surrogate for response (true vs. pseudoprogression, as measured with Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years (or up to 32 cycles) in the absence of disease progression or unacceptable toxicity. Patients also receive ferumoxytol IV and undergo MRI at baseline, 12 weeks after radiation, at suspected radiographic progression, and 6 weeks after suspected radiographic progression.

After completion of study treatment, patients are followed up at 30 days, every 12 weeks for up to 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have a histologically confirmed diagnosis of NSCLC
* Have up to ten measurable (by Response Assessment in Neuro-Oncology Criteria [RANO]) brain metastasis planned for stereotactic radiosurgery
* Have PD-L1 expression of greater than 1%
* Subjects may already be receiving PD-(L)1 (including pembrolizumab or other PD-[L]1 inhibitors such as nivolumab, atezolizumab, avelumab, durvalumab) for the treatment of systemic disease; a washout period of at least 3 weeks is required from the last dose of PD-(L)1 inhibitor
* Subjects with EGFR or ALK genomic tumor aberrations should have documented disease progression on Food and Drug Administration (FDA)-approved therapy for these aberrations; subjects with EGFR or ALK genomic tumor aberrations who develop new brain metastases may be included at the discretion of the treating physician
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin rime (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Has evidence of leptomeningeal disease on MRI or in cerebrospinal fluid (CSF)
* If tumor demonstrates EGFR or ALK genomic tumor aberrations, subject should have documented disease progression on FDA-approved therapy for these aberrations
* Has a diagnosis of immunodeficiency and is not on continuous daily immunosuppressive therapy within 7 days prior to the first dose of trial treatment; (subjects may receive steroids before or after SRS to prevent or manage cerebral edema; inhalational steroids are permitted)
* Has previously progressed on a PD-1 or PD-L1 checkpoint inhibitor for systemic disease
* Has a known history of active TB (Bacillus tuberculosis)
* Has hypersensitivity to pembrolizumab, gadolinium, or ferumoxytol or any of their excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier

  * Note: The use of denosumab is an exception to this criterion
* Subject who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: Subjects with =< grade 2 hematologic toxicities are an exception to this criterion and may qualify for the study
  * Note: Subjects with =< grade 2 fatigue are an exception to this criterion and may qualify for the study
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations; subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Subjects who have a contraindication for 3 tesla (3T) MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium containing contrast material
* Subjects with known iron overload (genetic hemochromatosis); in subjects with a family history of hemochromatosis, hemochromatosis must be ruled out prior to study entry with normal values of the following blood tests: transferrin saturation (TS) test and serum ferritin (SF) test; all associated costs will be paid by the study
* Subject who have received ferumoxytol within 3 weeks of study entry
* Subjects with three or more drug allergies from separate drug classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Relative Cerebral Blood Volume
Description: Will be analyzed using proportions and exact 95% confidence intervals. Sensitivity analysis will be based on subjects (lesions) with surgical results, and specificity analysis will be based on lesions with pseudo-progression determined based on surgical results or follow-up scan.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab When Given With Stereotactic Radiosurgery (SRS) in Subjects With Brain Metastasis
Description: Safety and tolerability will be determined using the Common Terminology Criteria for Adverse Events V4.0 (CTCAE) grades. They will be analyzed using percentages of patients who developed adverse events and exact 95% confidence intervals.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Best Response of Brain and Systematic Disease
Description: The duration of best response in brain and the duration of best response in systemic disease will be measured in months from the date on which criteria are met for complete response, partial response or stable disease until the first date that recurrent or progressive disease is objectively documented. Durations of best response will be analyzed using the Kaplan-Meier product limit estimates, taking censoring into account.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

4. Secondary Outcome: Best Response in Brain Disease
Description: Best response in brain disease will be measured based on brain MRI scan showing the best response to treatment and analyzed using proportions of categories of best response (e.g., complete remission, partial remission, progression, stable disease etc.) and exact 95% confidence intervals.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

5. Secondary Outcome: Best Response in Systematic Disease
Description: Best response in systematic disease will be measured based on body CT scan showing the best response to treatment and analyzed using proportions of categories of best response (e.g., complete remission, partial remission, progression, stable disease etc.) and exact 95% confidence intervals.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival will be measured in months from the date of diagnosis to the date of documented progression for each patient. Results will be analyzed using the Kaplan-Meier product limit estimates for all patients, taking censoring into account.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival will be measured in months from date of diagnosis to date of death. Results will be analyzed using the Kaplan-Meier product limit estimates for all patients, taking censoring into account.
Time Frame: Up to 2 years
Population: Due to low accrual and staffing issues, data was not collected for this outcome.
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse experiences will be recorded throughout the study and during the follow-up period (Up to 3 years).
Description: Adverse experiences will be graded and recorded according to NCI CTCAE Version 4.0. Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment
Arm/Group | Treatment (Pembrolizumab, Ferumoxytol MRI)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Ferumoxytol MRI) (N=2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Ferumoxytol MRI) (N=2)
Insomnia (Psychiatric disorders) | 1 (1)
Eye disorders- involuntary blinking (Eye disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb edema (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Elevated liver enzymes (Investigations) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to very low enrollment and staffing issues, data was not collected for analysis of study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03325166/Prot_SAP_000.pdf